CLINICAL TRIAL: NCT01868308
Title: Screening To Obviate Preterm Birth
Acronym: STOP
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 817085
Record Dates: First submitted 2013-05-29; First posted 2013-06-04 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Preterm Labor; Preterm Contractions; Abdominal Cramping; Back Pain; Vaginal Pressure; Vaginal Bleeding
MeSH Terms: conditions — Obstetric Labor, Premature; Colic; Back Pain; Uterine Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A vaginal swab will be collected during the patients clinical admission exam by a nurse.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Preterm Labor: Symptomatic women with singleton pregnancy at high risk for preterm birth between 22 - 33 6/7 weeks gestational age. We define "high risk for preterm birth" as women who present to our triage unit with complaints of preterm labor, including but not limited to preterm contractions, abdominal cramping, back pain, vaginal pressure, and vaginal bleeding.

SUMMARY:
Our objective is to investigate the predictive value of a panel of biomarkers associated with two biologically plausible pathways of preterm birth: membrane breakdown and cervical remodeling. The investigators will obtain cervical length, cervicovaginal fetal fibronectin, and a panel of novel cervicovaginal biomarkers associated with cervical remodeling in a prospective cohort of symptomatic women with a singleton pregnancy at high risk for preterm birth in an effort to better risk stratify this cohort.

DETAILED DESCRIPTION:
Preterm Birth is a complex syndrome for which several different biologically plausible pathways have been proposed, including mechanical uterine distension, abruption, inflammation, and/or activation of the fetal hypothalamic-pituitary-axis. However, despite our knowing the complexity of this syndrome and the different pathways involved, there is a paucity of clinical studies investigating whether detection of more than one of these pathways in a single patient might enhance the identification of those at greatest risk for preterm birth. We propose investigating the predictive value of a panel of biomarkers associated with two biological plausible pathways - membrane breakdown and cervical remodeling - that must be involved in the pathogenesis of preterm birth. Specifically, we propose measuring cervical length and collecting cervicovaginal fetal fibronectin as well as a panel of novel cervicovaginal biomarkers that reflect molecular pathways involved in cervical remodeling in a prospectively collected cohort of symptomatic women with singleton fetuses at high risk for preterm birth. Through this study we hope improve risk stratification of this high risk cohort.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy between 22- 33 6/7 weeks of gestational age.
* Must be experiencing one ore more of the following symptoms including but not limited to preterm contractions, abdominal cramping, back pain, vaginal pressure, or light vaginal bleeding.

Exclusion Criteria:

* Women with a multi-fetal pregnancy
* Intra uterine fetal demise
* Preterm premature rupture of membranes
* Overt chorioamnionitis

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All pregnant women presenting to the perinatal evaluation center at the Hospital of the University of Pennsylvania with preterm labor symptoms will be approached for the study.
Sampling Method: Non-Probability Sample
Enrollment: 589 (Actual)
Dates: Start 2013-01; Primary Completion 2015-02 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Preterm birth | Enrollment through delivery
  The primary outcome is preterm birth defined as delivery before 37 weeks.

SECONDARY OUTCOMES:
Early preterm birth | Enrollment through delivery
  The secondary outcome is "early" preterm birth defined as delivery before 34 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Michal A Elovitz, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States